CLINICAL TRIAL: NCT03149523
Title: Exhaustive Genetic and Immunological Characterization of Colon, Kidney and Liver Tumors to Define Potential Targets of Targeted and/or Immunomodulatory Therapies
Brief Title: Exhaustive Genetic and Immunological Characterization of Colon, Kidney and Liver Tumors
Acronym: ExhauCRF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: European Georges Pompidou Hospital (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Pierre Laurent-Puig, MD, PhD, European Georges Pompidou Hospital
Other Study IDs: CARPEM_ExhauCRF
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Adenocarcinoma; Hepatic Carcinoma; Kidney Adenocarcinoma
Keywords: exhaustive genetic and immunological analyses; targeted therapies; colon cancer; kidney cancer; liver cancer; immunological tumor microenvironment; tumor microenvironment heterogeneity
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Colonic Neoplasms; Kidney Neoplasms; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood samples, urine collection, tumor sample and tumor microenvironment sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Colorectal cancer: Patient with stage III colon carcinoma
- Kidney cancer: Patient with clear cell kidney carcinoma more than 4 cm surgically removed
- Liver cancer: Patient with advanced hepatocellular carcinoma : biopsy or resected BCLC (Barcelona Clinic Liver Cancer) stage B or C for diagnostic and/or therapeutic purposes

SUMMARY:
Over the last 10 years, technological advances in molecular biology enabled a more accurate genomic characterization of tumors. For each tumor location, this led to the identification of subgroups with similar molecular characteristics. This identification allowed the development of targeted therapies and thus to improve the patient prognosis. This molecular characterization has also revealed the tumor heterogeneity. It may be the cause of treatment resistance and therefore of relapses. Additionally, tumor cells are in constant dialogue with their microenvironment composed of different immune or non immune cells. This microenvironment is now targeted in cancer treatment.

To date, there are few studies that combine a deep genomic characterization of both tumor and tumor microenvironment of the patient. Combining the two types of studies on the same tumor should help to define new therapeutic targets and should allow a combination of targeted and immunomodulatory therapies. To this end, our project is to conduct an exhaustive integrated exploratory analysis at genomic, transcriptomic and immunological levels of 3 tumor types (in colon, kidney and liver cancer).

DETAILED DESCRIPTION:
The design consists in recruiting 50 patients per tumor location (colon, kidney, liver). For colorectal and kidney cancers, a prospective enrollment will be done for patients who have consented to the study. A retrospective enrollment will be done for patients with liver cancer only and who have consented to a national biological resource center form with genetic study approval.

The tumor samples will be taken during surgery. Blood and tumors samples will be taken as part of the treatment.

In case of a accidental germline discovery a management by a genetic consulting will be proposed.

ELIGIBILITY:
Inclusion Criteria:

* for colorectal cancer group : patient with stage III colon carcinoma
* for kidney cancer group : patient with primary clear cell carcinoma more than 4 cm
* for liver cancer group : patient with advanced hepatocellular carcinoma : biopsy or resected BCLC (Barcelona Clinic Liver Cancer) stage B or C
* patients who have consented to the study

Exclusion Criteria:

* Patients receiving neoadjuvant therapy are not eligible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal, kidney or liver cancers.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Sequencing of the exome and tumor RNA | Day of surgery
  Molecular classification of tumors

SECONDARY OUTCOMES:
HLA (human leukocyte antigen) typing | Day of surgery
  Prediction of neoantigens implicated in the intratumoral immune response
Immunophenotyping of intratumoral lymphocytes | Day of surgery
  Immunologic characteristic of tumors
Densities of lymphocytes T CD8 (cluster of differentiation 8) | Day of surgery
  Immunologic characteristic of tumors
Densities of macrophages M2 (CD68, CD163) | Day of surgery
  Immunologic characteristic of tumors
Densities of fibroblasts (SMA) | Day of surgery
  Immunologic characteristic of tumors
Quantification of lymphoid structures in immune infiltrate : DC-Lamp (Dendritic cell-lysosomal associated membrane protein)/CD3 | Day of surgery
  Immunologic characteristic of tumors
Quantification of lymphoid structures in immune infiltrate : CD20/CD3 | Day of surgery
  Immunologic characteristic of tumors
Expression profile of immune and stromal metagenes | Day of surgery
  Immunologic characteristic of tumors
Quantification of lymphocytes T CD4 (activated/inhibited) | Inclusion and 4 weeks after surgery
  Immunologic characteristic of circulating cells
Quantification of lymphocytes T CD8 (activated/inhibited) | Inclusion and 4 weeks after surgery
  Immunologic characteristic of circulating cells
Treg profile | Inclusion and 4 weeks after surgery
  Immunologic characteristic of circulating cells
MHC (major histocompatibility complex) peptide binding : Elispot | Inclusion and 4 weeks after surgery
  Immunologic characteristic of circulating cells
Cytokine assay : Luminex | Inclusion and 4 weeks after surgery
  Immunologic characteristic of circulating cells
Angiogenesis markers assay | Inclusion and 4 weeks after surgery
  Immunologic characteristic of circulating cells
Complement components assay | Inclusion and 4 weeks after surgery
  Immunologic characteristic of circulating cells
Transcriptomic profile of urinary RNAs | Inclusion
  Expression profile of immune gene in urine

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - AP-HP Jean Verdier Hospital, Bondy
  - AP-HP Cochin Hospital, Paris
  - AP-HP European Georges Pompidou Hospital, Paris

IPD SHARING:
Plan to Share IPD: No
The IPD (individual participant data) will not be shared. To protect confidentiality and integrity of patient information, only investigators of the study will have a regulated access to data with authorizations.